CLINICAL TRIAL: NCT02274337
Title: Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of AC0010 in Patients With Advanced Non Small Cell Lung Cancer Who Progressed on Prior Therapy With an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Agent
Brief Title: Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of AC0010 in Advanced Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Acea Bio (Hangzhou) Co., Ltd. (Industry); Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC0010-phaseI
Record Dates: First submitted 2014-10-19; First posted 2014-10-24 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Epidermal Growth Factor Receptor; Tyrosine Kinase Inhibitor; T790M mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AC0010 (Experimental): patients receiving avitinib treatment Qd, at different dose stages
  Interventions: Drug: AC0010

INTERVENTIONS:
Drug: AC0010 — patients take avitinib orally once per day at different dose

SUMMARY:
AC0010 Maleate Capsules is a new, irreversible, Epidermal Growth Factor Receptor (EGFR) mutation selective Tyrosine Kinase Inhibitor.Aim at local advanced or metastatic non-small cell lung cancer patients with EGFR mutation or T790M drug-resistant mutation. The molecular mechanism: by irreversible combining the EGFR-RTKs ATP binding site of cell, selectively suppress the activities of EGFR tyrosine kinase phosphorylation, block the sigal signal transduction system of EGFR, and close the function of ras/raf/MAPK downstream. at last block the tumor cell growth by EGFR induction, and promotes apoptosis. AC0010 Maleate Capsules has three characters: 1. Irreversible combination with EGFR; 2.Efficient suppress the EGFR mutant tumor cell and has no suppression to EGFR wild-type cell; 3. Efficient suppress the EGFR T790M drug-resistant mutation tumor cell.

DETAILED DESCRIPTION:
This study will treat patients with advanced NSCLC who have already received at least one course of specific anti-cancer treatment but the tumor has started to re-grow following that treatment. This is the first time that this drug is used or tested in patients, and so it will help to understand what type of side effects may occur with the drug treatment, it will measure the levels of drug in the body, it will also measure the anti-cancer activity. By using these pieces of information together the best dose of this drug to use in further clinical trials will be selected.

This study is a multicenter, open-label, two-stage phase I clinical trial. Trial including single-dose and successive-dose tolerance research, single-dose and successive-dose pharmacokinetic research, food bioavailability study, exploration of different dosing methods and tentative evaluation for clinical efficacy. Stage one is a dose escalation study, using the modified Fibonacci methods. 7 dose level are set, respectively are 50mg/d 100mg/d 200mg/d 350mg/d 550mg/d 850mg/d and 1100mg/d. Three patients are enrolled in each dose level, the observed indicator is dose-limited toxicity. No DLT occurred of all 3 patients, the dose escalate to next level. 1/3 DLT observed, 3 more patients are enrolled in the level, if no DLT is observed, the dose escalated to next level, if DLT occurs again, escalation stops. 2/3 DLT are observed, escalation stops. A recommend phase II dose level will acquire by this method. Stage two is a multicenter, open label, one arm successive dose clinical trial, based on the dosing level and method acquired in stage one, for further safety evaluation and tentative evaluation of clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender, aged from 18 years older to 70.
* Histologically or cytologically confirmed metastatic, or unresectable locally advanced, recurrent NSCLC.
* At least one measurable disease by CT or MRI, according to RECIST Version 1.1.
* Documented evidence of any activating EGFR mutation in the tumor tissue.
* Have undergone or are able to undergo a biopsy of either primary or metastatic tumor tissue within 28 days of dosing of Avitinib, and have tissue available to send to central lab for further genetic profiling especially the status of T790M.
* Life expectancy of at least 3 months.
* ECOG performance status of 0 to 1.
* Adequate hematological and physiological functions of heart, lung, liver, and kidney according to definitions given in Appendix D.
* Disease progression under at least one treatment with current marketed EGFR TKI therapy for at least 30 days (e.g. Erlotinib, or Gefitinib, or Afatinib) with intervening treatment after most recent EGFR TKI therapy. The washout period for an EGFR TKI (Erlotinib, or Gefitinib) is at a minimum of 7 days. The washout period for an irreversible EGFR inhibitor (Afatinib) and chemotherapy is at a minimum of 14 days.
* Any toxicity related to prior EGFR inhibitor treatment must have resolved to Grade 1 or less.
* NSCLC patients with asymptomatic brain metastasis or drug-controllable brain metastasis.
* Signed consent on an Independent Ethics Committee-approved Informed Consent Form prior to any study-specific evaluation.

Exclusion Criteria:

* No pathology confirmation
* History of interstitial lung disease related to prior EGFR inhibitor therapy.
* Symptomatic brain metastases or uncontrollable or unstable brain metastasis.
* Positive to HCV or HIV antibody.
* Treatment with prohibited medications (e.g., concurrent anticancer therapy including other chemotherapy, radiation, hormonal, or immunotherapy) ≤14 days prior to treatment with Avitinb.
* Clinically significant abnormal 12-lead ECG, QT interval corrected using Fridericia's method (QTcF) >450 msec (males) or >470 msec (females).
* Family history of long QT syndrome.
* Treatment with any Category 1 and 2 drugs (See:https://www.crediblemeds.org/ or www.qtdrug.org).
* Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study (e.g., substance abuse, uncontrolled psychiatric condition, uncontrolled intercurrent illness including active infection, arterial thrombosis, and symptomatic pulmonary embolism).
* Any other reasons for the investigator to consider the patient should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety, tolerability and ORR of AC0010 | Adverse events will be collected from baseline until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, ophthalmic examinations, RECIST1.1, and NCI CTCAE v4.03

SECONDARY OUTCOMES:
Plasma concentrations and pharmacokinetic parameters of single dose AC0010 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1 ,4 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48hours post dose)
  Plasma concentrations of AC0010 and 4 metabolites and pharmacokinetic parameters following single dose with fast in D1 and fed in D4 (Cmax, tmax, AUC, terminal rate constant, clearance, half life, volume of distribution and mean resistance time)
Plasma concentrations and pharmacokinetic parameters of multiple doses AC0010 | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 1, 8 ,15 and 22. D28- pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours post dose)
  Plasma concentrations of AC0010 and 4 metabolites and pharmacokinetic parameters following multiple doses (steady state Cmax, tmax, Cmin AUC, clearance, accumulation ratio and time dependency)
Efficacy of AC0010 | CT or MRI at screening and every 4-8 weeks (from first dose of multiple dosing) until disease progression or withdrawal from study, expected average 6 months
  Evaluation of tumour response, duration of response, tumour shrinkage, progression free survival and overall survival as assessed by RECIST 1.1
Food effect on AC0010's bioavailibility | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 4 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48hours post dose)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China